CLINICAL TRIAL: NCT04960111
Title: Radiostereometry (Model Based RSA) in the Assessment of Knee Prosthesis Outcome:a Prospective,Pilot,Single-center Study.
Brief Title: Radiostereometry in Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RSA
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Knee Osteoarthritis; Knee Arthropathy; Aseptic Loosening
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- knee arthroplasty with radiostereometry tecnique (Experimental): patient underwent total knee arthroplasty with insertion of microsphere in tantallium for radiostereometry tecnique.
  Interventions: Device: RSA

INTERVENTIONS:
Device: RSA — application of tantalium microsphere around knee prosthesis and RSA X-ray post operative to detect early mobilization in follow up.

SUMMARY:
The innovative aspect of this research is the possibility of combining the data collected with radiostereometric model based Radiostereometry with the data collected through the Galeazzi Institute Registry.This opens the prospect of an earlier identification of patients undergoing prosthetic knee replacement with initial aseptic loosening.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18
* patients underwent total knee arthroplasty without controindications for this procedure
* patients enrolled in PatientsReportedOutcomesMeasureS (PROMS) study

Exclusion Criteria:

* age less than 18
* comorbility that make difficult come back for follow-up
* patients with allergy at materials used in Radiostereometry tecnique
* infection
* anemia, obesity, osteoporosis
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-07-10 (Estimated)

PRIMARY OUTCOMES:
micro-movement detection with radiostereometry and the patient's perception, measured with Short Form health survey12 at 12 month after surgery. | 12 months
  evaluate correlation between levels of micro-movement of the prosthetic components using radiostereometry model based RSA and the patient's perception, measured with Short Form health survey12 at 12 month after surgery.

SECONDARY OUTCOMES:
correlation of micromovements and Patient reported outcomes at follow up | baseline to 24 months
  evaluate correlation between levels of micro-movement of the prosthetic components using radiostereometry model based RSA and the patient's perception, measured with patient reported oucomes used in Galeazzi Institute Registry at each post operative follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided